CLINICAL TRIAL: NCT00821106
Title: Transradial Approach [LEft vs Right] aNd Procedural Times During Percutaneous Coronary Procedures: TALENT Study
Brief Title: Left Versus Right Transradial Approach for Percutaneous Coronary Procedures
Acronym: TALENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Casilino ASL RMB (Other)
Responsible Party: Alessandro Sciahbasi MD, UOC Cardiologia-Policlinico Casilino-ASL RMB-Rome-Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TALENT
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-01

CONDITIONS: Coronary Angiography; Angioplasty, Transluminal, Percutaneous Coronary
Keywords: Coronary angiography; percutaneous coronary intervention; Transradial approach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right transradial approach (Experimental): Coronary diagnostic or interventional procedures performed through right radial approach
  Interventions: Procedure: Right radial
- Left transradial approach (Experimental): Diagnostic or interventional procedures performed through left radial approach
  Interventions: Procedure: left radial

INTERVENTIONS:
Procedure: Right radial — diagnostic or interventional procedures performed through right transradial approach
  Arms: Right transradial approach
Procedure: left radial — diagnostic or interventional procedures performed through left transradial approach
  Arms: Left transradial approach

SUMMARY:
Transradial approach of cardiac catheterization is a common alternative to transfemoral access for diagnostic coronary angiography and percutaneous coronary interventions (PCI). The transradial approach reduces access site bleeding complications and the procedural discomfort of the patients. Transradial procedures may be performed by cannulation of the right or left radial artery and at present, the choice of the right or left radial artery depends largely on the operator' s preference.

The aim of this study is to evaluate safety and efficacy of transradial approach comparing the right radial versus the left radial approach in coronary diagnostic and interventional procedures.

The investigators will enroll consecutively for 12 months all patients who undergo to diagnostic or interventional procedures through trans radial approach in two Italian centers (Casilino Policlinic, Catholic University-Rome).

Primary end point of the study is the fluoroscopy time and the radiation dose adsorbed by the patients. Secondary end-points are: contrast amount, time to obtain the first angiography, procedural shift rate, number of catheters employed, major complications.

The investigators pre-specified a sub-study in patients older than 75 years old with the same end-points.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo to diagnostic or interventional procedures

Exclusion Criteria:

* Previous coronary artery by-pass
* Acute myocardial infarction with ST segment elevation myocardial infarction
* Cardiogenic shock
* Ischemic Allen Test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1540 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Primary end point of the study is the fluoroscopy time of the procedure and the radiation dose adsorbed by the patients | 7 days

SECONDARY OUTCOMES:
Contrast amount, time to obtain the first angiography, procedural shift rate, number of catheters employed, major complications. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sciahbasi, MD, Principal Investigator — Policlinico Casilino ASL RMB
Locations (2):
- Italy (2):
  - Policlinico Casilino-ASL RMB, Rome
  - Università Cattolica del Sacro Cuore, Rome